CLINICAL TRIAL: NCT00448292
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy of PRX-00023 in Patients With Major Depressive Disorder.
Brief Title: A Efficacy Study of PRX-00023 in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epix Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPX-CP-020
Record Dates: First submitted 2007-03-13; First posted 2007-03-16 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Depression; Major Depressive Disorder; Major Depression; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — naluzotan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PRX-00023 taken twice daily, escalating from 40 mg to 80 mg to 120 mg
  Interventions: Drug: PRX-00023
- 2 (Placebo Comparator): Placebo taken twice daily, escalating from 40 mg to 80 mg to 120 mg
  Interventions: Drug: Placebo for PRX-00023

INTERVENTIONS:
Drug: PRX-00023 — Doses taken two times per day. dose increased at scheduled intervals from 40 mg to 80 mg to 120 mg.
  Arms: 1
Drug: Placebo for PRX-00023 — Doses taken two times per day. dose increased at scheduled intervals from 40 mg to 80 mg to 120 mg.
  Arms: 2

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled study is to assess the safety and efficacy of PRX-00023 in patients with major depressive disorder.

DETAILED DESCRIPTION:
Patients with major depressive disorder who meet all of the eligibility criteria will be randomly assigned to receive twice daily doses of either placebo or PRX-00023. Study drug will be taken for up to approximately 9 weeks. Patients will have periodic office visits for the purpose of monitoring safety and tolerability, as well as efficacy assessments.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of major depressive disorder

Key Exclusion Criteria:

* Females who are pregnant or nursing
* Electroconvulsive therapy within previous year
* Type 1 diabetes or uncontrolled type 2 diabetes
* HIV, Hepatitis B or Hepatitis C
* Use of illegal drugs, history of drug abuse, and/or alcohol dependence
* Clinically significant abnormal lab results

Other protocol-defined eligibility criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2007-03; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Montgomery-Asberg Depression Rating Scale (MADRS). | change from baseline through end of study

SECONDARY OUTCOMES:
Side effects during and immediately following the treatment period | assessed throughout study
changes from baseline on the Hamilton Anxiety Rating (HAM-A) scale | change from baseline through end of study
changes from baseline on the Quick Inventory of Depressive Symptomatology-self report (QIDS-SR) | change from baseline through end of study
changes from baseline on the Clinical Global Impressions (CGI) scale | change from baseline through end of study
responder and remission rates | change from baseline through end of study
changes from baseline on the Changes in Sexual Function (CSFQ) scale. | change from baseline through end of study

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Vista Medical Research, Inc., Mesa, Arizona
  - Pharmacology Research Institute, Encino, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Synergy Clinical Research Center, National City, California
  - Excell Research, Oceanside, California
  - Pacific Clinical Research Medical Group, Riverside, California
  - AVI Clinical Research, Torrance, California
  - Pacific Clinical Research Medical Group, Upland, California
  - GWU Clinical Psychiatric Research Center, Washington D.C., District of Columbia
  - CNS Healthcare of Jacksonville, Jacksonville, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Chicago Research Center, Inc., Chicago, Illinois
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Brentwood Research Institute, Shreveport, Louisiana
  - Piedmont Neuropsychiatry, Charlotte, North Carolina
  - University of Pennsylvannia, Philadelphia, Pennsylvania
  - SE Health Consultants, LLC, Charleston, South Carolina
  - University of Texas - Southwestern Medical Center, Dallas, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network, Seattle, Washington